CLINICAL TRIAL: NCT04009733
Title: Epigenetic Regulation of Osteogenesis Imperfecta Severity : miROI Study
Acronym: miROI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL19_0021; 2019-A00521-56 (Other: ID-RCB)
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2023-05

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis imperfecta; micro Ribonucleic acids; epigenetics
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Osteogenesis imperfecta type 1 (Experimental): Patients with OI type 1
  Interventions: Biological: Blood sample
- Osteogenesis imperfecta type 3 (Experimental): Patients with OI type 3
  Interventions: Biological: Blood sample
- Control population (Active Comparator): The control population corresponds to a pre-existing serum collection of osteoarthritis cohorts (OFELY and MODAM for women, STRAMBO for men).
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — A study specific blood sample will be collected.
  Arms: Osteogenesis imperfecta type 1; Osteogenesis imperfecta type 3
Biological: Blood sample — Pre-collected serum of cohort OFELY and MODAM for women, STRAMBO for men will be used for the study.
  Arms: Control population

SUMMARY:
Osteogenesis Imperfecta (OI) is a heterogeneous group of rare connective tissue hereditary diseases responsible for fragility and bone deformity. OI is caused by an autosomal dominant mutation of COL1A1 or COL1A2, encoding α1 and α2 of the collagen, regardless of their phenotypic severity (1 to 5 OI type).

This observation suggests the existence of a undetermined mechanism that may be found in epigenetic regulation, including particularly micro Ribonucleic Acids (miRs).

Indeed, these small non-coding miRs are involved in the regulation of major steps of cellular processes in different pathologies, especially in bone disease.

Currently, no study can provide a satisfactory answer.

This is an etiologic study to reveal the correlation between micro-RNAs (miR) expression and the type I or III of the Osteogenesis Imperfecta (OI).

The aim of this study is therefore to identify miRs significantly associated with the severity of OI.

ELIGIBILITY:
Inclusion Criteria:

Control population:

* Male or female
* 18 years old and over
* Be part of cohorts STRAMBO, OFELY or MODAM

Patients with OI:

* Male or female ≥18 years old
* Have COL1A1 or COL1A2 mutation
* Have a diagnosis of type 1 or 3 from Silence classification made by a rheumatologist expert in bone pathologies

Exclusion Criteria:

* Refusal to participate in the study
* Have received glucocorticoid treatment for more than 3 months
* Have received anti-osteoporotic treatment for less than 1 year ago
* Have Chronic inflammatory rheumatism
* Have an uncontrolled hypo/hyper thyroidism ou hypo/hyper parathyroidism
* Have cancer or bone metastases (current or in the past two years)
* Have benign bone tumors or Paget's disease
* Have malabsorptive disease (Celiac disease, Whipple's disease, intestinal bypass, short bowel syndrome) and inflammatory bowel disease
* Pregnant or lactating women
* Have psychiatric disorders seriously hindering understanding
* Have difficulties in oral understanding of French language
* Not a beneficiary of french social security
* Patients protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2022-04-24 (Actual)

PRIMARY OUTCOMES:
micro Ribonucleic Acids (miRs) expression in serum of the patients Osteogenesis imperfecta (OI) type I or III versus control population | up to 1 month (after inclusion)
  Identification of specific miRs expressed in the serum of OI patients using NGS (Next Generation Sequencing).

SECONDARY OUTCOMES:
Nature of micro Ribonucleic Acids (miRs) identified by Next-Gen Sequencing (NGS ) | Up to 1 month (after inclusion)
  Compare the nature of the miRs identified by NGS (Next Generation Sequencing) in serum between the 3 groups of subjects: type 1 Osteogenesis Imperfecta (OI), type 3 OI and controls (controls are patients with osteoarthritis).
Level of expression of micro Ribonucleic Acids (miRs) identified by Next-Gen Sequencing (NGS ) | Up to 1 month (after inclusion)
  The objective is to validate expression of miRs identified by NGS (Next Generation Sequencing) in blood samples of patients from 3 groups: an Osteogenesis imperfecta (OI) type 1 cohort and an OI type 3 cohort, recruited for the study, and a pre-existing group of control patients (issued from cohorts OFELY and MODAM for women, STRAMBO for men).
  Expression of the significant miRs identified by NGS will be measured by Reverse Transcription Quantitative Polymerase Chain Reaction (RT-qPCR) and then these results will be compared with same analysis on blood samples of control patients.
Presence of fracture | Up to 1 month (after inclusion)
  Severity of OI will be evaluated using radiological data (fracture) extracted from patients' medical records. Association between expression of miRs in patients with OI with the severity of the disease will be studied by statistical analysis.
Presence of biochemical markers of bone turnover in blood | Up to 1 month (after inclusion)
  Severity of OI will be evaluated using biological data (biochemical markers of bone turnover) extracted from patients' medical records. Association between expression of miRs in patients with OI with the severity of the disease will be studied by statistical analysis.
Bone pain | Up to 1 month (after inclusion)
  Severity of OI will be evaluated using clinical data (bone pain mesured on Visual Analogue Scale) extracted from patients' medical records. Association between expression of miRs in patients with OI with the severity of the disease will be studied by statistical analysis.
Quality of life | Up to 1 month (after inclusion)
  Investigators will use a specific questionnaire completed by a rheumatologist at inclusion to obtain more information about a patient's lifestyle. The higher the score the more severe the disease impact and vice versa. Association between expression of miRs in patients with OI with the severity of the disease will be studied by statistical analysis.
Assessment of environmental factors | Up to 1 month (after inclusion)
  The investigating team will use information extracted from patients' medical records to obtain environmental information, which includes using a specific questionnaire completed by a rheumatologist with patients at inclusion.
  Association between expression of miRs in patients with OI with the environmental data will be studied by statistics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Roland CHAPURLAT, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Result] Mercier-Guery A, Millet M, Merle B, Collet C, Bagouet F, Borel O, Sornay-Rendu E, Szulc P, Vignot E, Gensburger D, Fontanges E, Croset M, Chapurlat R. Dysregulation of MicroRNAs in Adult Osteogenesis Imperfecta: The miROI Study. J Bone Miner Res. 2023 Nov;38(11):1665-1678. doi: 10.1002/jbmr.4912. Epub 2023 Oct 2. PMID 37715362